CLINICAL TRIAL: NCT03613909
Title: Acceptance of the CP950 Sound Processor With Experienced CP810/CP910/CP920 BTE Sound Processor Users
Brief Title: Acceptance of the CP950 Sound Processor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLTD5591
Record Dates: First submitted 2016-01-31; First posted 2018-08-03 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Hearing Loss, Sensorineural
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Intervention Model Description: Repeated measures, single-subject experiment. Each subject received the same treatment.
Oversight: Data Monitoring Committee: No

ARMS (1):
- All participants (Experimental): At least 6 months experience with a Nucleus 24 series or later implant in at least one implanted ear and at least 3 months experience with the CP810,CP920 or CP910 sound processor.
  Interventions: Device: CP950 OTE Sound processor

INTERVENTIONS:
Device: CP950 OTE Sound processor — CP950 is Off The Ear (OTE) Cochlear Implant Sound Processor

SUMMARY:
Acceptance of CP950 sound processor with experienced CP810/CP910/CP920 BTE sound processor users.

ELIGIBILITY:
Inclusion Criteria:

1. Eighteen years of age or older
2. At least 6 months experience with a Nucleus 24 series or later implant in at least one implanted ear
3. At least 3 months experience with the CP810,CP920 or CP910 sound processor
4. Native speaker in the language used to assess speech perception performance
5. Willingness to participate in and to comply with all requirements of the protocol
6. Able to score 30% or more at +15 SNR with CI alone

Exclusion Criteria:

1. Unrealistic expectations on the part of the subject, regarding the possible benefits, risks and limitations that are inherent to the procedure and prosthetic device
2. Additional disabilities that would prevent participation in evaluations
3. Nucleus 22 Implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Protocol stated "up to 25" number of participants. 23 were enrolled, with 3 electing to withdraw from the study before completion.
Period: First Take Home Use of CP950
Arm/Group | All Participants
Started | 23
Completed | 20
Not Completed | 3
Period: First In Booth Testing of CP950
Arm/Group | All Participants
Started | 20
Completed | 20
Not Completed | 0
Period: Second Take Home Use of CP950
Arm/Group | All Participants
Started | 20
Completed | 20
Not Completed | 0
Period: Second In Booth Testing of CP950
Arm/Group | All Participants
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All Study Participants
Groups:
- All Participants: All participants enrolled in the study
Arm/Group | All Participants
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 7
Age, Continuous [Mean (Full Range); unit: years] | 57 [30 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Australia | 23

OUTCOME MEASURES:

1. Primary Outcome: Acceptability Ratings for the CP950 Sound Processor Compared to Subjects' Own Processors, Summarized by the Overall Hearing Performance Score.
Description: Each subject used the Investigational device (CP950) for take home use to obtain subjective ratings.
  During the take home use, A subjective questionnaire was asked them to recall and rate how their hearing performance with the Investigational device CP950 OTE processor compared to their hearing performance with their own CP810, CP910 or CP920 BTE processor.
  Likert scale was used for each rating in the questionnaire for at home usage ( with the values ranging from) : 1 = much worse; 2 = somewhat worse; 3 = No difference; 4 = somewhat better; 5 = much better.
Time Frame: 14 days
Measure: Mean (Inter-Quartile Range); unit: Units on a likert scale
Arm/Group | All Participants
Number analyzed (Participants) | 20
Units on a likert scale | 3.6 [2 to 5]

2. Secondary Outcome: Speech Reception Threshold (SNR50) for Sentence Testing in Noise With CP950 Sound Processor .
Description: Signal to noise ratio (measured in decibels) providing 50% speech intelligibility for sentences presented in noise to evaluate the benefit from microphone directionality with the CP950 OTE (Off the ear) sound processor.
Time Frame: in booth testing 1 day.
Measure: Mean (Standard Error); unit: decibles
Arm/Group | All Participants
Number analyzed (Participants) | 20
decibles | 4 (0.5)

3. Secondary Outcome: Percentage of Correct Words Scored With Sentences in Noise With the CP950 Sound Processor
Description: Two lists of twenty sentences presented from front speaker with 4 Talker babble noise presented from rear-half speakers. Higher the percentage of correct words means better outcome.
Time Frame: In booth testing 1 day
Measure: Mean (Standard Deviation); unit: percentage of correct words.
Arm/Group | All Participants
Number analyzed (Participants) | 20
percentage of correct words. | 49.82 (3.9)

ADVERSE EVENTS:
Time Frame: 11 months
Description: Adverse events were collected during the periods when participants were using the investigational device (CP950).
Groups:
- All Participants: At least 6 months experience with a Nucleus 24 series or later implant in at least one implanted ear and at least 3 months experience with the CP810, CP920 or CP910 sound processor.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 19/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=20)
Discomfort Headache and pain (Investigations) | 9 (9) — Discomfort/pain/headache at the site of the processor magnet.
Tinnitus (Ear and labyrinth disorders) | 2 (2)
Loud Crackling sound (Ear and labyrinth disorders) | 1 (1)
Vertigo and pre planned hospitalization (General disorders) | 3 (3)
Ear infection (Infections and infestations) | 1 (1)
Fall at car park (Social circumstances) | 1 (1)
Pain at the site of processor magnet (Investigations) | 1 (1)
Pleurisy (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes